CLINICAL TRIAL: NCT05383560
Title: Phase 2, Randomized, Observer-Blind, Investigator-Initiated, Collaborative Study to Evaluate the Safety and Immunogenicity of Omicron Variant-Matched Vaccine Booster in Adults
Brief Title: Safety and Immunogenicity of Omicron Variant-Matched Vaccine Booster in Adults
Acronym: SH-MO-214
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Principal Investigator, Gili Regev-Yochay MD, Director of Infection Prevention & Control Unit, Sheba Medical Center
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: Sheba-22-9312
Record Dates: First submitted 2022-05-15; First posted 2022-05-20 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: COVID-19 Pandemic; Immunogenicity; SARS CoV 2 Infection; COVID-19
Keywords: mRNA1273.214; Omicron; Immunogenicity; COVID-19; Safety; mRNA1273.222
MeSH Terms: conditions — COVID-19 | interventions — mRNA-1273.214 COVID-19 vaccine; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Intervention Model Description: Protocol versions 1.01-1.06:Randomized, Observer-Blinded (2:2:1 ratio) Protocol version 1.07:Randomized, Observer-Blinded (1:1 ratio)
Who Masked: Participant, Investigator
Masking Description: Pharmacy will be responsible for all IPs masking, using a masking sleeve on ready to use each injection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- mRNA-1273.214 + mRNA-1273.214 (Experimental): Fourth & Fifth doses of an investigational mRNA vaccine, 56 days apart N ≈ 60 Under protocol versions 1.01-1.06
  Interventions: Biological: mRNA-1273.214 Vaccine
- mRNA-1273.214 + Placebo (Experimental): Fourth dose of an investigational mRNA vaccine followed by a fifth dose of placebo, 56 days apart N ≈ 60 Under protocol versions 1.01-1.06
  Interventions: Biological: mRNA-1273.214 Vaccine; Biological: Placebo
- mRNA-1273 + Placebo (Active Comparator): Fourth dose of the commercial mRNA vaccine, followed by a fifth dose of placebo, 56 days apart N ≈ 30 Under protocol versions 1.01-1.06
  Interventions: Biological: MRNA-1273 Vaccine; Biological: Placebo
- mRNA-1273.214 (Experimental): A booster dose of an investigational mRNA vaccine at Visit 1 (Day 1). N ≈ 30 Under protocol versions 1.07
  Interventions: Biological: mRNA-1273.214 Vaccine
- mRNA-1273.222 (Active Comparator): A booster dose of the commercial mRNA vaccine at Visit 1 (Day 1). N ≈ 30 Under protocol versions 1.07
  Interventions: Biological: MRNA-1273.222 Vaccine

INTERVENTIONS:
Biological: mRNA-1273.214 Vaccine — Omicron Variant-Matched Vaccine
  Arms: mRNA-1273.214; mRNA-1273.214 + Placebo; mRNA-1273.214 + mRNA-1273.214
Biological: MRNA-1273 Vaccine — Moderna's commercial COVID-19 Vaccine
  Other Names: Spikevax
  Arms: mRNA-1273 + Placebo
Biological: Placebo — Normal Saline for injection
  Arms: mRNA-1273 + Placebo; mRNA-1273.214 + Placebo
Biological: MRNA-1273.222 Vaccine — Moderna's commercial COVID-19 Vaccine
  Other Names: Spikevax Bivalent
  Arms: mRNA-1273.222

SUMMARY:
Under protocol versions 1.01-1.06: The five recently emerged SARS-CoV2 variants that were designated as VOCs are the Alpha variant, Beta variant, Gamma variant, Delta variant and the Omicron variant. The current dominant Omicron variant was designated a VOC by WHO on Nov 26, 2021, and was found to comprise 85% of reported variants in late January 2022. Studies have shown that the prevalent Omicron mutations in the S1 subunit RBD region and NTD region could dramatically change the antigenic features of the viral spike, leading to significantly reduced neutralization Omicron harbors 30 signature mutations (>50% prevalence) of which 15 are in the S1 subunit RBD region and 8 are in the S1 subunit NTD region. Omicron is a highly contagious variant with threatening immune evasion capabilities even despite robust immune response. Initial modeling showed the Omicron variant being 2.8 times more infectious than the Delta variant. While current vaccines are losing protection against Omicron with respect to infection and mild disease, there is still considerable protection from hospitalisation and severe COVID-19, especially after a booster dose. The International Coalition of Medicines Regulatory Authorities (ICMRA) COVID-19 Omicron Variant Workshop encouraged the international scientific community and vaccine developers to look at alternative approaches to monovalent vaccines. In ICMRA's view, companies should also explore the feasibility of developing bivalent or multivalent variant vaccines to determine if they offer advantages to monovalent vaccines. As advised by ICMRA, the investigated vaccine, mRNA-1273.214 is a bivalent vaccine containing the ancestral SARS-CoV-2 and the Omicron variant spike sequences that will be evaluated as a heterologous boost.

Under protocol version 1.07:The study will also investigate the safety, reactogenicity and immune response of the mRNA-1273.222 administered as a boost vaccine after primary series vaccination comprising 3 doses of an mRNA vaccine .

This study hypothesizes that the peak level of antibodies against SARS CoV-2, will be at two weeks after the first study dose is administered, which is similar to other recent findings (Anderson et al., 2022).2.2.1. The bivalent mRNA-1273.222 vaccine contains mRNA encoding for the spike protein of BA.4/BA.5 as well as mRNA encoding for the original (ancestral Wuhan-Hu-1) strain of the SARS-CoV-2 virus.

DETAILED DESCRIPTION:
Under protocol versions 1.01-1.06:The trial aims to evaluate the safety and immunogenicity of the investigated covalent vaccine, mRNA-1273.214, administered as a heterologous vaccine after the primary series vaccination and boost with the BNT162b2 or mRNA-1273, in healthy adults aged ≥21 years.

Three different treatment arms will be compared with participants being administered either:

1. mRNA-1273.214 (Day 1) and mRNA-1273.214 (Day 56)
2. mRNA-1273.214 (Day 1) and placebo (Day 56)
3. mRNA-1273 (Day 1) and placebo (Day 56)

Study procedures include two administrations of vaccine and/or placebo, nasopharyngeal swab for SARS-CoV-2 PCR, blood draws for antibody response: IgG, IgA, pseudo-neutralization antibody (ab) titers, B-Cell response, T-Cell response, and solicited and non-solicited adverse events. Subjects will be asked to complete an electronic diary for 7 consecutive days after each vaccination dose, regarding vaccine-related symptoms + temperature measured at home. One week after the day of vaccination or placebo, subjects will be asked to complete a COVID-19 questionnaire once a week, in which they will have to answer the question of whether they have experienced COVID-19 symptoms. Adverse reactions will be measured by the occurrence of solicited injection site reaction and systemic reaction from the time of each vaccination through 7 days post each vaccination/placebo administration. Unsolicited non-serious Adverse Events (AEs), Serious adverse events (SAEs), new-onset chronic medical conditions (NOCMCs), and medically-attended adverse events (MAAEs) will be collected from baseline through 6 months after the first booster dose vaccination.

Nasopharyngeal Swab for SARS-CoV-2 PCR, Blood Samples For Immunogenicity Assessment, Serology and PBMC will be collected at each study visit (6 times during the subject's participation in the study).

Under protocol version 1.07:The trial aims is to evaluate the safety and immunogenicity of the messenger-RNA (mRNA) based bivalent vaccine candidates mRNA-1273.214 and mRNA-1273.222 administered as second and/or third boosts to healthy adults aged ≥25 years who received at least a primary series of 3 doses of mRNA vaccination. The total study population will include 180 subjects.

The study will include two (2) additional arms. At Visit 1 (Day 1), subjects will be administered a booster dose of mRNA-1273.222 vaccine (arm 4), or mRNA-1273.214 vaccine (arm 5). Up to 60 subjects will be enrolled for arms 4 and 5 (~30 subjects per arm).

Note: all subjects enrolled under protocol versions 1.01-1.06 (arms 1-3) will continue with their planned procedures as described in protocol version 1.06.

Subjects enrolled under protocol version 1.07 (arms 4 and 5), will participate in five (5) visits:

Visit 1 (Day 1) Visit 2 (Day 15 ± 3 days) Visit 3 (Day 29 + 12 days) Visit 4 (Day 91 ± 7 days) Visit 5 (Day 181 ± 14 days) The injection with the investigated vaccine booster mRNA-1273.214 (Arm 4) or mRNA-1273.222 (Arm 5) will be given at Visit 1.

Unblinding for subjects enrolled under protocol version 1.07 will be performed at Visit 4 (Day 91 ± 7 days).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 21 years of age, inclusively.
2. Protocol versions 1.01-1.06:Individuals who previously received mRNA primary series vaccination AND a booster dose at least 4 months prior to Day 1. Documented confirmation of prior mRNA series vaccination receipt must be obtained prior to randomization. Protocol version 1.07:Individuals who had previously received mRNA primary series vaccination comprising at least 3 vaccine doses with the last one at least 6 months prior to Day 1. Documented confirmation of prior mRNA series vaccination receipt must be obtained prior to randomization. Note: subjects who had received 4 vaccine doses (i.e., a primary series of 3 doses and an additional boost) may also be enrolled under protocol version 1.07).
3. Females and males of childbearing potential must be willing to use effective methods of contraception such as hormones (OCP, oral contraceptive pill), condom or occlusive cap with spermicidal agents, intrauterine device (IUD), or intrauterine system (IUS) as well as to refrain from donating sperm through 28 days following the last vaccination.
4. Participant who is willing and able to comply with all scheduled visits, vaccination plan, laboratory tests, lifestyle considerations, and other study procedures.
5. For Women of Child Bearing Potential (WOCBP): a negative pregnancy test on the day of vaccination (Visit 1 and Visit 4).
6. Participant who is willing and able to operate an electronic diary.
7. Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.

   Note: Healthy participants with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the six (6) weeks before enrollment, can be included.
8. Capable of giving signed informed consent as described which includes understanding and compliance with the study procedures, requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
9. Must agree not to enroll in another study of an investigational agent prior to completion of the study.

Exclusion Criteria:

1. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (e.g., anaphylaxis) to any component of the study intervention(s).
2. Previous clinical (based on COVID-19 symptoms/signs alone, if a SARS-CoV-2 NAAT result was not available) or microbiological (based on COVID-19 symptoms/signs and a positive SARS-CoV-2 NAAT result) diagnosis of COVID-19 or positive antigen test for SARS-CoV-2 at baseline.
3. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
4. Has known or suspected allergy or history of anaphylaxis, urticaria, or other significant AR to the vaccine or its excipients.
5. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
6. Inability to observe possible local reactions at the injection sites due to a physical condition or permanent body art.
7. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
8. Pregnant or breastfeeding women.
9. Individuals who receive treatment with radiotherapy or immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids (if systemic corticosteroids are administered for ≥14 days at a dose of ≥20 mg/day of prednisone or equivalent), e.g., for cancer or an autoimmune disease, or planned receipt throughout the study. Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
10. Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days before study intervention administration, or receipt of any passive antibody therapy specific to COVID-19, from 90 days before study intervention administration, or planned receipt throughout the study.
11. Participation in other studies involving study intervention within 28 days prior to study entry through and including 28 days after the last dose of study intervention.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Safety of the study vaccines after each dose | 6 Months
  Safety of the study vaccines will be measured by solicited and unsolicited adverse injection site reactions and systemic reactions from the time of each vaccination through 7 days post each vaccination/placebo administrations. AEs will be collected up to 29 days after injection. Unsolicited non-serious AEs, SAEs, NOCMCs, and MAAEs will be collected through 6 months after the first vaccine dose.
Reactogenicity of the study vaccines after each dose | 6 Months
  Reactogenicity of the study vaccines will be measured by solicited and unsolicited adverse injection site reactions and systemic reactions from the time of each vaccination through 7 days post each vaccination/placebo administrations. AEs will be collected up to 29 days after injection. Unsolicited non-serious AEs, SAEs, NOCMCs, and MAAEs will be collected through 6 months after the first vaccine dose. The study will also assess reactogenicity using "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials" Guide, via an electronic diary the participants would be required to complete every day for 7 consecutive days starting the day of each vaccine.
Immune response to mRNA-1273.214, given as a fourth and fifth dose to participants who previously received mRNA primary series vaccination and one booster dose (third dose). | 6 Months
  Primary immunogenicity outcome will be measured by changes in geometric titers (GMTs) and geometric fold raise (GMFRs) of IgG and neutralizing antibodies (nAb), using a pseudovirus assay during all visits. Blood for immunogenicity will be collected at all visits (total of 6 visits).

SECONDARY OUTCOMES:
Immunogenicity | 6 Months
  Describe direct virus neutralization of Omicron VOC, Delta VOC and ancestral SARS-COV-2 VOC. Direct virus neutralization (in Biosafety Level 3 - BL3 - facility) of Omicron variant of concern (VOC) and two (2) additional strains [ancestral SARS-COV-2 and Delta VOC] Measured by GMT.
Investigational Product's Efficacy | 6 Months
  COVID-19 infections and severity [based on CDC definition] in participants without evidence of past SARS-CoV-2 infection, occurring after day 7 from the booster dose throughout the blinded follow-up period. Laboratory defined SARS-CoV-2 infection and symptomatic COVID-19 and severe COVID-19.

OTHER OUTCOMES:
Exploratory Immunogenicity | 6 Months
  Under protocols versions 1.01-1.06: Characterize T-cell activation post-boost 1273.214, Interferon Gamma per 106 cells. Characterize B-cell responses post-boost 1273.214. IgA response (IgA GMTs). Characterize any breakthrough cases of SARS-CoV-2 infections or COVID-19 and any SARS-CoV-2 isolates by Culture isolates for optional sequencing.
  Under protocol version 1.07: Characterize T-cell activation post-boost 1273.214 or post-boost 1273.222. Characterize B-cell responses post-boost 1273.214 or post-boost 1273.222 and assessment of IgA response.
Describe the immune response to mRNA-1273.214 and mRNA-1273.222 by assessment of Changes in Neutralizing Antibodies. | Under protocol version 1.07: 6 Months
  Blood samples will be collected for the assessment of Changes in Neutralizing Antibodies from Visit 1 to Visit 3, and Visit 5.
Describe the immune response to mRNA-1273.214 and mRNA-1273.222 by Comparison of Neutralizing Antibodies against SARS-CoV-2 Wild Type and newly emerged variants | Under protocol version 1.07: 6 Months
  Blood samples will be collected for the Comparison of Neutralizing Antibodies against SARS-CoV-2 Wild Type and newly emerged variants in Arm 4 (mRNA-1273.214) vs. Arm 5 (mRNA-1273.222) at Day 29 (Visit 3) and Day 181 (Visit 5).
COVID-19 infections (based on CDC definition) in subjects without evidence of past SARS-CoV-2 infection, occurring after day 7 from the booster dose throughout the blinded follow-up period. | Under protocol version 1.07: 6 Months
  Will be measure in the following lab tests: nasopharyngeal swab for SARS-CoV-2 polymerase chain reaction (PCR) test and antigen test. A positive result of antigen test will require SARS-CoV-2 polymerase chain reaction test to confirm COVID-19 infection.
COVID-19 severity in subjects without evidence of past SARS-CoV-2 infection, occurring after day 7 from the booster dose throughout the blinded follow-up period. | Under protocol version 1.07: 6 Months
  Will be measure according to the COVID-19 symptoms that will be reported by the subjects and graded according to the CTCAE V 5.0 or if occurred during the first 7 days after receiving vaccine boost, according to the Adverse Reaction Grading Scale (Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. 2007).

CONTACTS AND LOCATIONS:
Overall Officials: Gili Regev-Yochay, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes
Unidentified data will be available after publication of the results.
Supporting Information: Study Protocol, SAP
Time Frame: will be available upon publication of results
Access Criteria: Upon request. Requires collaborator's approval as well.

REFERENCES:
- [Derived] Lustig Y, Barda N, Weiss-Ottolenghi Y, Indenbaum V, Margalit I, Asraf K, Doolman R, Chalkias S, Das R, Elfatarany G, Harats D, Kreiss Y, Regev-Yochay G. Humoral response superiority of the monovalent XBB.1.5 over the bivalent BA.1 and BA.5 mRNA COVID-19 vaccines. Vaccine. 2024 Sep 17;42(22):126010. doi: 10.1016/j.vaccine.2024.05.058. Epub 2024 May 27. PMID 38806352